CLINICAL TRIAL: NCT03603431
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose-escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Activity of MRG-110 Following Local Intradermal Injection After Skin Excisional Wound Creation in Normal Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MRG-110 Following Intradermal Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MRG110-01-001
Record Dates: First submitted 2018-07-09; First posted 2018-07-27 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteers; MicroRNAs; Angiogenesis Inducing Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose - MRG-110 (Experimental): Intradermal injection of MRG-110 at two wound sites and intradermal injection of placebo at two other wound sites
  Interventions: Drug: MRG-110; Drug: Placebo
- Single Ascending Dose - Placebo (Placebo Comparator): Intradermal injection of placebo at four wound sites
  Interventions: Drug: Placebo
- Multiple Ascending Dose - MRG-110 (Experimental): Intradermal injection of MRG-110 at two wound sites and intradermal injection of placebo at two other wound sites
  Interventions: Drug: MRG-110; Drug: Placebo
- Multiple Ascending Dose - Placebo (Placebo Comparator): Intradermal injection of placebo at four wound sites
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MRG-110 — Single ascending doses of MRG-110
  Arms: Single Ascending Dose - MRG-110
Drug: Placebo — Single doses of placebo
  Arms: Single Ascending Dose - MRG-110; Single Ascending Dose - Placebo
Drug: MRG-110 — Multiple ascending doses of MRG-110
  Arms: Multiple Ascending Dose - MRG-110
Drug: Placebo — Multiple doses of Placebo
  Arms: Multiple Ascending Dose - MRG-110; Multiple Ascending Dose - Placebo

SUMMARY:
MRG-110 is intended to promote the growth of new blood vessels by inhibiting a molecule called miR-92a. MRG-110 is being studied to determine if it can accelerate healing of wounds by improving blood flow into the wound area. The primary objective of this study is to investigate the safety and tolerability of MRG-110 when injected into the skin at the site of a small skin wound in normal healthy volunteers. Another objective is to study the pharmacokinetics of MRG-110 (the movement of a drug into, through and out of the body). Participants in the clinical trial will receive either a single dose or multiple doses of MRG-110 and/or placebo. Blood samples, urine samples and skin biopsies will be collected to measure how MRG-110 is processed by the body, and how the body responds when exposed to MRG-110.

ELIGIBILITY:
Key Inclusion Criteria:

* Normal healthy volunteers.
* Females must be of non-childbearing potential.
* If engaged in sexual relations with a female of child-bearing potential, males must be surgically sterile or must be willing to use a highly effective method of contraception throughout their study participation and for at least 6 months after the last dose of study drug.
* Must have 2 regions on lower back/upper buttocks that are free of striae, scars, tattoos, or other skin pathologies.
* Must have no conditions that could increase risk of abnormal or delayed healing.

Key Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical examination.
* Clinically significant abnormalities in laboratory tests at screening.
* History of cutaneous disorder.
* Hemangioma, history of hemangioblastoma, or other known vascular disorder.
* Positive for bloodborne pathogen (hepatitis B, hepatitis C, HIV).
* Use of an investigational drug or device within 28 days prior to Day 1, or use of an investigational biological or oligonucleotide drug within 90 days of Day 1.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | Up to Day 55

SECONDARY OUTCOMES:
Area under the plasma concentration vs. time curve (AUC) of MRG-110 following single and repeat doses. | Up to Day 45
Peak plasma concentration (Cmax) of MRG-110 following single and repeat doses | Up to Day 45

OTHER OUTCOMES:
Area of granulation tissue formation | Day 11 or Day 18
Histological markers of angiogenesis (such as CD31, ERG, ITGA5) | Day 11 or Day 18
Wound perfusion measured by laser speckle imaging | Up to Day 45
Proportion of wounds closed over time | Up to Day 55

CONTACTS AND LOCATIONS:
Overall Officials: Diana Escolar, MD, Study Director — miRagen Therapeutics, Inc.
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Huang CK, Kafert-Kasting S, Thum T. Preclinical and Clinical Development of Noncoding RNA Therapeutics for Cardiovascular Disease. Circ Res. 2020 Feb 28;126(5):663-678. doi: 10.1161/CIRCRESAHA.119.315856. Epub 2020 Feb 27. PMID 32105576